CLINICAL TRIAL: NCT06540937
Title: Phase II Clinical Study of Leflunomide in the Treatment of MEN-1 Neuroendocrine Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2409
Record Dates: First submitted 2023-02-18; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Neuroendocrine Tumors
Keywords: Multiple Endocrine Neoplasia; Leflunomide
MeSH Terms: conditions — Neuroendocrine Tumors; Multiple Endocrine Neoplasia | interventions — Leflunomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leflunomide tablets (20 mg orally, once a day, before going to bed) were administered every 28 days (Experimental): Eligible patients will receive leflunomide tablets (20 mg orally, once a day, before bed) every 28 days until the disease progresses or adverse reactions become intolerable.
  Interventions: Drug: Leflunomide Pill

INTERVENTIONS:
Drug: Leflunomide Pill — This is a single-arm, single-center, phase II clinical study. Primarily evaluated in advanced MEN-1 neuroendocrine tumors. The initial efficacy of leflunomide tablets in second-line treatment provided evidence for phase III clinical trials.
  Other Names: Leflunomide 20mg

SUMMARY:
This phase II trial studies aim to evaluate the initial efficacy of leflunomide tablets in second-line treatment of advanced MEN-1 neuroendocrine tumors, and to provide evidence for phase III clinical trials.

DETAILED DESCRIPTION:
1. Treatment methods Eligible patients will receive leflunomide tablets (20 mg orally, once a day, before bed) every 28 days until the disease progresses or adverse reactions become intolerable.
2. Follow-up Eligible patients should follow the requirements of the study protocol and continue to the end of the study. The purpose of the follow-up is to know whether the subjects have adverse reactions to the treatment effect and take appropriate treatment. Evaluation should be conducted every two cycles. If the test is terminated before disease progression, the subjects should be followed up every 6 weeks for imaging examination to observe whether the tumor progresses. Other antitumor therapy, hepatotoxic drugs (phenylbutazone, phenytoin, methotrexate, methyldopa, rifampicin) and traditional Chinese medicine were not allowed before the group withdrawal.

   At each follow-up, the patient's history is taken, and the following examinations are performed: physical examination; Blood routine, urine routine, liver and kidney function, serum tumor markers, electrocardiogram; Tumor imaging (e.g., chest and abdominal CT); Blood biomarker test; other tests required for the condition.
3. Tumor tissue/blood biomarker examination In this project, the mutation of MEN-1 gene of the patient should be tested, and blood samples of the patient and tumor tissue samples remaining during routine diagnosis and treatment should be collected. The remaining samples will be returned to the Cancer Hospital of Chinese Academy of Medical Sciences for storage. The results of these tests will determine whether the patient can participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, gender unlimited
* Pathological diagnosis of neuroendocrine tumor
* MEN-1 germ line mutation (MEN-1 syndrome), or tumor with somatic MEN-1 mutation
* Unresectable neuroendocrine tumors that have failed standard first-line systemic therapy
* At least one evaluable lesion according to the RECIST criteria
* ECOG physical condition score: 0-1
* Voluntarily joined the study, signed the informed consent, complied well, and cooperated with the follow-up.
* Must meet the following requirements: Bone marrow: leukocyte > 4.0×109/L, neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥10g/dL; Liver: total bilirubin < 1.5 times the upper limit of normal, AST/ALT≤1.5 times the upper limit of normal value, Lactate dehydrogenase ≤1.5 times the upper limit of normal value, Alkaline phosphatase ≤5 times the upper limit of normal value; Kidney: serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance ≥60ml/min

Exclusion Criteria:

* Received any antitumor therapy within 4 weeks
* Participated in or are participating in clinical trials of other drugs/therapies within 4 weeks prior to the initial use of the study drug
* Underwent/received major surgery or has not recovered from the side effects of the surgery within 4 weeks prior to the initial use of the study drug
* Subjects of other malignant tumors unless complete remission was achieved at least 2 years prior to study inclusion and not required other treatment during the study period
* Persistent or active (serious) infection
* Hypertension that is difficult to control with medication (continuous blood pressure is greater than 150/90 MMHG
* Poorly controlled diabetes
* Grade II/IV congestive heart failure or heart block
* Within 6 months prior to use for the first time seen in the following situations:

Deep vein thrombosis; Pulmonary embolism; Myocardial infarction; Serious arrhythmia; Instability or angina pectoris; Percutaneous coronary intervention; Acute coronary syndrome; Coronary artery bypass grafting

* Be allergic to leflunomide tablets and their metabolites
* Severe liver damage
* Other severe acute or chronic medical conditions or abnormalities in laboratory tests that may increase the risks associated with study participation or may interfere with the interpretation of study results
* Poor compliance, or other conditions unsuitable for participation in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by RECIST 1.1 | up to 36 weeks
  ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) according to RECIST v1.1.
Progression-free survival (PFS) | up to 36 weeks
  PFS is defined as the duration from the date of randomization to the onset of tumor progression or death of any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 36 weeks
  OS is defined as the time from the date of randomization until death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhao, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma Y, Zhu Q, Wang X, Liu M, Chen Q, Jiang L, Chi Y, Zeng YX, Zhao H, Jiao Y. Synthetic lethal screening identifies DHODH as a target for MEN1-mutated tumor cells. Cell Res. 2022 Jun;32(6):596-599. doi: 10.1038/s41422-022-00613-1. Epub 2022 Feb 15. No abstract available. PMID 35169281